CLINICAL TRIAL: NCT01910467
Title: Avoiding Hypotension in Preterm Neonates (AHIP) - A Randomised Controlled Study on Near Infrared Spectroscopy Monitoring of Peripheral-muscle and Cerebral Oxygenation With Defined Interventions Versus Routine Monitoring and Treatment in Preterm Neonates
Brief Title: Avoiding Hypotension in Preterm Neonates
Acronym: AHIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pichler Gerhard, MD., Ass. Prof. Dr., Medical University of Graz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15351
Record Dates: First submitted 2013-07-19; First posted 2013-07-29 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIRS visible and predefined interventions (Experimental): NIRS measurements are visible and the patients will be treated according to predefined clinical interventions: If cTOI/pTOI ratio increases >5% within a six-hours-period echocardiography will be performed and based on results of echocardiography and blood pressure a volume bolus or, if ventilated, modification of ventilation or treatment of patent ductus arteriosus will be considered.
  Interventions: Device: NIRS visible and predefined interventions
- NIRS not visible and treatment as usual (Other): NIRS measurements are not visible and the patients will be treated according to routine ('treatment as usual')
  Interventions: Device: NIRS not visible and treatment as usual

INTERVENTIONS:
Device: NIRS visible and predefined interventions — NIRS measurements are visible and the patients will be treated according to predefined clinical interventions: If cTOI/pTOI ratio increases >5% within a six-hours-period echocardiography will be performed and based on results of echocardiography and blood pressure a volume bolus or, if ventilated, modification of ventilation or treatment of patent ductus arteriosus will be considered.
  Arms: NIRS visible and predefined interventions
Device: NIRS not visible and treatment as usual — NIRS not visible and the patients will be treated according to routine
  Arms: NIRS not visible and treatment as usual

SUMMARY:
Objectives Firstly to examine in preterm neonates, whether it is possible to reduce number of hypotensive episodes and use of catecholamines by applying cerebral/peripheral near infrared spectroscopy in combination with predefined interventions and secondly to explore the potential impact on cerebral injury and mortality.

Hypothesis By using predefined interventions for changes in cerebral/peripheral oxygenation ratio investigators will reduce hypotensive episodes and use of catecholamines which will reduce cerebral injury and mortality.

Methods Cerebral (cTOI) and peripheral-muscle (pTOI) tissue-oxygenation-index (NIRO 300) will be measured for 24h starting <6 hours postpartum. When cTOI/pTOI ratio increases >5% within a 6h period, predefined interventions will be performed.

Primary outcome parameter will be duration of hypotensive episodes and use of catecholamines during the first 48h after birth. Secondary outcome parameters will be cerebral injury and mortality.

ELIGIBILITY:
Inclusion Criteria:

* preterm neonates
* decision to conduct full life support
* written informed consent
* age <6 hours
* no use of catecholamines before start of NIRS measurements

Exclusion Criteria:

* no decision to conduct full life support
* no written informed consent
* age >6 hours
* use of catecholamines before start of NIRS measurements
* congenital malformation

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2013-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time (percentage of hours) of hypotension/use of catecholamines during the first 48 hours | 48 hours

SECONDARY OUTCOMES:
Cerebral injury by cerebral ultrasound | up to 16 weeks
  From date of randomization until the date of discharge or date of 40 weeks of gestational age, whichever came first, assessed up to 16 weeks.
Mortality | up to 16 weeks

OTHER OUTCOMES:
Neonatal morbidities | up to 16 weeks
  From date of randomization until the date of discharge or date of 40 weeks of gestational age, whichever came first, assessed up to 16 weeks.
Heart rate | 48 hours
Blood pressure | 48 hours
Arterial oxygen saturation | 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, MD, Principal Investigator — Dep. of Pediatrics, Medical University of Graz
Locations (1):
- Dep. of Pediatrics, Medical University of Graz, Graz, Styria, Austria

REFERENCES:
- [Derived] Hoeller N, Baik-Schneditz N, Schwaberger B, Mileder L, Urlesberger B, Pichler G. Cerebral and peripheral muscle oxygenation and perfusion: Course in moderate and late preterm neonates during the first day after birth. Physiol Int. 2020 Jul 17;107(2):267-279. doi: 10.1556/2060.2020.00028. PMID 32692715
- [Derived] Pichler G, Holler N, Baik-Schneditz N, Schwaberger B, Mileder L, Stadler J, Avian A, Pansy J, Urlesberger B. Avoiding Arterial Hypotension in Preterm Neonates (AHIP)-A Single Center Randomised Controlled Study Investigating Simultaneous Near Infrared Spectroscopy Measurements of Cerebral and Peripheral Regional Tissue Oxygenation and Dedicated Interventions. Front Pediatr. 2018 Feb 1;6:15. doi: 10.3389/fped.2018.00015. eCollection 2018. PMID 29450194